CLINICAL TRIAL: NCT07065071
Title: Mentalization-Based Therapy (MBT) With Older Adults: A Hermeneutic Single-Case Efficacy Design (HSCED) Series
Brief Title: Mentalization-Based Therpay With Older Adults
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Derbyshire Healthcare NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 24072; 349077 (Other: IRAS Project ID)
Record Dates: First submitted 2025-03-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-02

CONDITIONS: Mentalisation; Mentalization; Later Life; Older Adults; Attachment; Borderline Personality Disorder
Keywords: mentalisation; mentalization; later life; older adults; attachment trauma; borderline personality disorder; attachment; bpd; mbt; mentalisation-based therapy; mentalization-based therapy
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Mentalization-Based Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Older adults: People aged 60+ who are eligible for Derbyshire Healthcare NHS Foundation Trust's Later Life MBT group
  Interventions: Other: Mentalization-Based Therapy

INTERVENTIONS:
Other: Mentalization-Based Therapy — Group MBT that takes place as part of treatment as usual within Derbyshire Healthcare NHS Foundation Trust's Older Adult Community Mental Health Team's service.
  Other Names: MBT; Mentalisation-Based Therapy

SUMMARY:
The investigators would like to find out if Mentalization-Based Therapy (MBT) is effective for people aged 60+ who struggle in relationships. The study aims to understand whether MBT helps older people to build better relationships and feel better about themselves. There is currently no research with people over 60 and MBT, yet MBT is being offered to the older adult population by NHS trusts throughout the UK without evidence for its effectiveness. As well as developing knowledge about how MBT can help at this point in life, the study aims to improve the quality of care offered.

MBT targets mentalization, which is the ability to make sense of one's own and other people's thoughts, feelings, actions and beliefs. Current research suggests that the ability to mentalize changes over the lifespan and may be influenced by many factors, some of which are specific to later life. For example, changes in relationships during later life and biological changes in the brain may impact mentalization systems.

The investigators would also like to understand what difficulties MBT may be effective for in later life. The diagnosis of borderline personality disorder (BPD), which MBT was developed to treat, was, until recently, assumed to disappear with age. However, growing evidence suggests that symptoms change, rather than disappear.

Given these unknowns, the study will use a Hermeneutic Single-Case Efficacy Design (HSCED). Up to six participants, up to six people who know the participants, and clinicians delivering the MBT interventions will be recruited. Data in the form of questionnaires, self-report and therapy documents will be gathered, and everyone will be interviewed. For each participant, the data will be used to compile both an affirmative (yes, MBT was effective) case, and a sceptic case (no, MBT was not effective). Cases will then be reviewed by an adjudication panel comprising one service user expert by experience, one MBT expert and one expert in another therapeutic modality. For each case, each expert will decide if the affirmative or sceptic case was more likely. Finally, findings will be synthesised and used to draw conclusions about the effectiveness of MBT.

The HSCED lends itself to theory-building, as it gathers in-depth data from individuals and facilitates comparison within and between cases. Further, participants' contribution to their own 'rich case record' through change interviews recognises people as taking an active role in their own healing.

DETAILED DESCRIPTION:
Study Design The study will involve single-centre convenience-sampling recruitment from a Later Life MBT Group run within Older Adult Community Mental Health Teams (CMHT) within Derbyshire Healthcare NHS Foundation Trust. The MBT intervention groups have been established for approximately 12 months and constitute an existing referral pathway within the Older Adult CMHT service. Given this, the study takes an observational design, as although participants receive a therapeutic intervention (MBT) the investigators will not assign a specific intervention to participants, rather they will recruit participants from an already established MBT group. The MBT intervention that participants will be receiving is therefore 'treatment as usual'.

The study will use a Hermeneutic Single-Case Efficacy Design (HSCED), an interpretative framework for evaluating causality between processes and outcomes in psychotherapeutic interventions (Elliott, 2001; Elliott, 2002). Based on several of Wall et al.'s (2017) HSCED adaptations, the study will recruit four to six participants (depending on drop-out rate), informants (people who know the participants), and four clinicians delivering the MBT intervention. This will allow for case-wise comparison and provide greater evidence for considering efficacy theory. Data collected will be both quantitative (questionnaires) and qualitative (free-form questionnaires, therapy documents and interviews).

Affirmative and sceptic cases will be developed and reviewed by the research team to ensure a fair presentation of the data. In addition, the HSCED design limits bias by the inclusion of the adjudicational panel, comprising judges who are independent of the research team. One judge will be an expert in MBT, one an expert in another therapeutic modality, and the final judge will be a service user who identifies as an older adult with attachment difficulties, offering the perspective of someone who might be eligible for the MBT intervention. For each participant, each expert will decide if the affirmative or sceptic case was more likely. Finally, findings will then be synthesised and used to draw conclusions about the effectiveness of MBT.

ELIGIBILITY:
Inclusion Criteria:

Participants - people who:

* Have been referred into and assessed as suitable for a Derbyshire Healthcare NHS Foundation Trust's Later Life MBT Group
* Have persistent (i.e. 1 year+) and pervasive (i.e. multiple relationships) difficulties in relationships and so stand to benefit from the intervention
* Those aged 60+
* Have the ability to complete measures
* Can communicate comfortably in spoken and written English

Informants - people who:

* Are identified by the participant
* Are aged 18+
* The participant considers themselves to have a close relationship with
* Have the ability to complete appropriate measures
* Can communicate comfortably in spoken and written English

Clinicians - people who:

• Are involved in delivering/facilitating the MBT interventions with participants

Exclusion Criteria:

Participants - people who:

* Are undertaking any other psychological intervention
* Do not have the capacity to give informed consent; since capacity is dynamic, this will be assessed by clinicians and the independent outcome assessor on an ongoing basis according to their clinical judgement. If lack of capacity is identified during an interview, clinical judgement would be used around rescheduling and the information would be fed back to the individual's clinical team or escalated as necessary

Informants - people who:

• Do not have the capacity to give informed consent; since capacity is dynamic, this will be assessed by the independent outcome assessor according to their clinical judgement. If lack of capacity was identified during an interview, clinical judgement would be used around rescheduling and the information would be escalated as necessary

Clinicians - people who:

• n/a

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to six participants will be recruited via purposive convenience sampling from people enrolled on one of Derbyshire Healthcare Foundation Trust's (DHCFT's) Later Life MBT interventions. The MBT group interventions take place in a secondary care outpatient setting.
  Once participants have been recruited, they will be asked to invite someone with whom they have a close relationship to participate in the study, known as the informant. Up to six informants will be recruited in this way via purposive convenience sampling.
  Up to four clinicians running the Later Life MBT intervention will be recruited via purposive convenience sampling, since they will be the people already running the group.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder 7-item questionnaire (GAD-7) | Administered at baseline, the end of the introduction to MBT phase (roughly 7 weeks), and 6 months subsequent to this.
  The GAD-7 is a self-report measure of 7 questions pertaining to frequency of symptoms of anxiety experienced over the past 2 weeks. Responses are given on a Likert scale ranging from 0-3, where 0 = 'not at all' and 3 = 'nearly every day', with higher scores indicating greater severity of symptoms of anxiety. Administered to participants.
Personal Health Questionnaire, 9-item (PHQ-9) | Administered at baseline, the end of the introduction to MBT phase (roughly 7 weeks), and 6 months subsequent to this.
  The PHQ-9 is a self-report measure of 9 questions pertaining to frequency of symptoms of depression experienced over the past 2 weeks. Responses are given on a Likert scale ranging from 0-3, where 0 = 'not at all' and 3 = 'nearly every day', with higher scores indicating greater severity of symptoms of depression. Administered to participants.
Recovering Quality of Life 10 (ReQoL-10) | Administered at baseline, the end of the introduction to MBT phase (roughly 7 weeks), and 6 months subsequent to this. Also administered weekly at the start of MBT sessions for the duration of the MBT intervention (6 months and 7 weeks).
  The ReQoL-10 is a self-report measure of 10 questions pertaining to the respondent's frequency of thoughts, feelings and activities relevant to quality of life over the last week. Responses are given on a Likert scale ranging from 0-4, where 0 = 'none of the time' and 4 = 'most or all of the time', with higher scale scores indicating higher quality of life. Administered to participants.
Certainty About Mental States Questionnaire (CAMSQ) | Administered at baseline, the end of the introduction to MBT phase (roughly 7 weeks), and 6 months subsequent to this. Also administered weekly at the end of MBT sessions for the duration of the MBT intervention (6 months and 7 weeks).
  The CAMSQ is a self-report measure of 20 questions exploring respondent's interpretations of the thoughts, feelings and behaviours of themselves and others. Responses are given on a Likert scale ranging from 0-6, where 0 = 'never' and 6 = 'always'. For scoring, items are divided into two subscales, Certainty about Self and Certainty about Others. High scores on Self-Certainty and middling scores on Other-Certainty are considered to reflect adaptive mentalizing. Administered to participants.
Brief Reflective Functioning Interview (BRFI; adapted) | Administered at baseline, the end of the introduction to MBT phase (roughly 7 weeks), and 6 months subsequent to this.
  The Brief Reflective Functioning Interview (BRFI) is a short semi-standardized interview that is based on the Adult Attachment Interview (AAI), in which participants are asked to reflect on any relationship with someone they have known for a long time. This adapted version is based on Rudden (2010). There are 9 questions, including 'Can you tell me about a specific memory with that person from when you were younger that shows something about your relationship?' and 'Why did you choose to speak about this person?'. Administered to participants. Responses will be coded using the Reflective Functioning Scale to ascertain levels of mentalizing.
Helpful Aspects of Therapy Questionnaire (HAT) | Administered weekly at the end of MBT sessions for the duration of the MBT intervention (6 months and 7 weeks).
  The HAT is a qualitative self-report measure of 7 questions exploring helpful and hindering events during therapy sessions. Respondents are asked to briefly write their answers to questions such as 'Of the events which occurred during this session, which one do you feel was the most helpful or important for you personally?', 'Did anything happen during the session that might have been hindering?', 'About where in the session did this event occur?' and 'How long did this event last?'. Respondents are also invited to quantitatively rate the helpfulness of the event using a Likert scale ranging from 1-9, where 1 = 'extremely hindering' and 9 = 'extremely helpful'. Administered to participants and clinicians.
Mentalization-Based Therapy (MBT) Adherence & Competence Scale | Administered weekly at the end of MBT sessions for the duration of the MBT intervention (6 months and 7 weeks).
  The MBT Adherence & Competence Scale is a self-report measure of 18 items pertaining to fidelity to the MBT model. Ratings are given on a Likert scale ranging from 0-7, where 0 = 'not at all' and 7= 'extensively', where higher scores indicate higher fidelity to MBT. The scale accounts for Frequency, Extensiveness and Quality of interventions, including whether an intervention is absent when it should have been used. Completed by clinicians.
Change Interview Schedule | Administered at the end of the introduction to MBT phase (roughly 7 weeks), and 6 months subsequent to this.
  The Change Interview Schedule is a semi-structured interview schedule exploring change, adapted from Elliot (1996) and Elliot (1999). There are 11 questions including 'What has the MBT group been like for you (so far)?' and 'In general, what do you attribute these various changes to? In other words, what do you think might have brought them about? Both outside and inside of being in the group.' Administered to participants, informants and clinicians.
MBT Documents | Administered at the end of the introduction to MBT phase (roughly 7 weeks), and 6 months subsequent to this.
  Any documents or paperwork completed or created by participants during MBT will be analysed for change over time and/or themes related to mentalization.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schröder, PhD, Study Director — University of Nottingham; Heather Cogger-Ward, DClinPsy, Principal Investigator — University of Nottingham; Helen Philpott, DClinPsy, Study Director — Derbyshire Healthcare NHS Foundation Trust; Laura Hayward, DClinPsy, Study Director — Derbyshire Healthcare NHS Foundation Trust
Locations (1):
- Derbyshire Healthcare NHS Foundation Trust, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided